CLINICAL TRIAL: NCT05448833
Title: V-Lap System For Wirelessly Measuring And Monitoring Left Atrial Pressure (Lap) In Patients With Advanced Chronic Heart Failure
Brief Title: V-Lap System For Wirelessly Measuring And Monitoring Left Atrial Pressure (LAP) In Patients With Advance Chronic Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vectorious Medical Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLC-0021
Record Dates: First submitted 2022-06-26; First posted 2022-07-07 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- V-LAP™ System (Experimental): Heart failure subjects - Percutaneous implantation of the V-LAP™ implant by right heart catheterization (RHC) approach and daily LAP measurements at home and will be trained on the use of the device for self-management.
  Interventions: Device: V-LAP™ SYSTEM

INTERVENTIONS:
Device: V-LAP™ SYSTEM — Delivery of the V-LAP™ implant by right heart catheterization. A catheter-based approach in a trans-septal puncture procedure, deploying it in the inter-atrial septum.

SUMMARY:
The objective of this study is to evaluate the safety and performance of the V-LAP System in subjects with New York Heart Association (NYHA) functional class II and III HF, irrespective of left ventricular ejection fraction.

DETAILED DESCRIPTION:
The trial is designed to demonstrate that the V-LAP™ implant can be positioned in the interatrial septum.

The V- LAP™ System is intended for wirelessly measuring and monitoring LAP. The V-LAP™ System is indicated for subjects with chronic symptomatic ACC/AHA Stage C.

Pressure-guided medical management of study participants, with the goal of reducing hospitalizations and improving quality of life, will be implemented using a physician-directed patient self-management approach.

V-LAP-PSM (Patient Self-management), Patient Guidance Application is a smartphone application that guides the patient on how to self-adjust the treatment, according to physician prescription, and when to approach the study investigator.

Safety will be monitored by the occurrence of adverse events throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

- 1. Ischemic or non-ischemic cardiomyopathy and documented heart failure for at least 6 months (diagnosis of HF ≥ 6 months), regardless of ejection fraction.

2. NYHA Class II heart failure (HF) subjects, documented at Baseline Visit regardless of ejection fraction, meeting both inclusion criteria in subsections (2a) and (2b) or NYHA Class III heart failure (HF) subjects, documented at Baseline Visit regardless of ejection fraction, meeting at least one inclusion criteria in subsections (2a) and (2b).

1. Have a minimum of one (1) HF hospitalization or equivalent (HF Emergency Department Visit or HF Urgent Clinic Visit) within the last 12 months associated with signs/symptoms of congestion requiring treatment with intravenous (IV) diuretic. If Cardiac Resynchronization Therapy (CRT) device previously implanted, the HF hospitalization or equivalent must be ≥ 30 days after CRT implantation.
2. Have a corrected* elevated outpatient Brain Natriuretic Peptide (BNP) level of at least 300 pg/ml or an N-terminal pro-BNP (NT-proBNP) level of at least 1,500 pg/ml, according to local measurement, within 90-days of the Baseline Visit.

   *Thresholds for NT-proBNP will be corrected for body mass index (BMI) using a 4% reduction per BMI unit over 20 kg/m2. If subject is on ARNI, NT-proBNP should be used exclusively.

   3. Receiving maximally-tolerated medical therapy for heart failure as indicated per ACC/AHA or ESC Heart Failure Guidelines (guideline-directed medical therapy or GDMT), in the absence of contraindications and lack of availability. GDMT refers to those guideline-directed medical therapies having a Class I indication for use.
   * For patient with heart failure and a reduced ejection fraction (HFrEF), GDMT includes a diuretic as needed for volume control, angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) or angiotensin receptor neprilysin inhibitor (ARNI), beta-blocker (BB), mineralocorticoid receptor antagonist (MRA), and SGLT2 inhibitor for at least 3 months prior to the Baseline visit. Drug doses, with the exception of diuretics, should be stable for at least 1 month, where stability is defined as no more than a 100% increase or 50% decrease in dose.
   * For patient with heart failure and a preserved ejection fraction (HFpEF), GDMT includes a diuretic as needed for volume control and treatment of associated conditions (e.g., hypertension, atrial fibrillation) for at least 3 months prior to the Baseline visit. Drug doses, with the exception of diuretics, should be stable for at least 1 month, where stability is defined as no more than a 100% increase or 50% decrease in dose.
   * Patients should also receive Class I recommended cardiac rhythm management device therapy. Specifically: if indicated by class I guidelines, cardiac resynchronization therapy (CRT), implanted cardioverter-defibrillator (ICD), or a pacemaker should be implanted at least 3 months prior to Baseline Visit. These criteria may be waived if a patient is clinically contraindicated for these therapies or refuses them and must be attested to by the investigator.
   * GDMT may change over time; the most current versions of the ACC/AHA or ESC Heart Failure Guidelines will supersede the above guidelines.

     4. Provide informed consent for study participation and be willing and able to comply with the required tests, treatment instructions, and follow-up visits.

   Exclusion Criteria:
   * 1. Age less than 22 (<22) or greater than 88 (>88) years old. 2. Subjects who are NYHA class IV and ACC/AHA stage D. 3. Subjects with evidence/history of a major cardiovascular or neurovascular event, such as an intra-cardiac thrombus or history of stroke, transient ischemic attack, systemic or pulmonary thromboembolism, deep vein thrombosis (DVT), within the last 6 months of Baseline Visit.

     4. Subjects with a resting systolic blood pressure <90 or >180 mmHg. 5. Left ventricular end-diastolic diameter (LVEDD) > 8cm. 6. Have an atrial septal defect or patent foramen ovale with more than trace shunting on color Doppler or intravenous bubble study or surgical or interventional correction of congenital heart disease involving atrial septum, including placement of a PFO or ASD closure device, and have a hypermobile septum or a septal aneurysm.

     7. Subjects with untreated severe valve lesions, which are indicated for surgical or percutaneous intervention, active valvular vegetations, atrial myxoma, hypertrophic cardiomyopathy with significant resting or provoked subaortic gradient, acute myocarditis, tamponade, or large pericardial effusion, constrictive pericarditis, infiltrative cardiomyopathy (including cardiac sarcoidosis, amyloidosis, and hemochromatosis), or congenital heart disease, as a cause of HF.

     8. Uncontrolled tachyarrhythmia or bradycardia (heart rate <45). 9. Intractable HF with resting symptoms despite maximal medical therapy (ACC/AHA HF Stage D), including subjects receiving continuous or intermittent outpatient IV vasoactive medications (e.g., IV inotropes, IV vasodilators), subjects treated with a ventricular assist device (VAD).

     10. Intolerant to ACE-I, ARB, or ARNI and beta-blocker medical therapy for subjects classified as HFrEF (EF ≤40%).

     11. The presence of an acute coronary syndrome (ACS), percutaneous coronary intervention (PCI), rhythm management system revision, lead extraction, or cardiac or other major surgery within the preceding 90 days.

     12. Subjects not eligible for emergency open-heart, thoracic or vascular surgery.

     13. Women of childbearing age. 14. Subjects with a life expectancy that is shorter than 12 months, or those who have received a cardiac transplant or are listed for cardiac transplantation and likely to be transplanted within 12 months of Baseline Visit.

     15. Have coagulopathy or uninterruptible anticoagulation therapy or contraindication for all the forms of antiplatelet/anticoagulant treatments anticipated in the protocol.

     16. Known history of life-threatening allergy to contrast dye that cannot be properly pre-medicated.

     17. Have an estimated Glomerular Filtration Rate (GFR) <20 ml/min/1.73 m2 by the MDRD method or on chronic renal dialysis.

     18. Hepatic impairment with at least one liver Function Test (transaminases, total bilirubin, or alkaline phosphatase) ≥ 3 times upper limit of normal.

     19. Gastrointestinal bleeding in the last 6 months. 20. Have severe chronic pulmonary disease requiring continuous home oxygen, chronic oral steroid therapy, hospitalization for exacerbation during prior 6 months, or has severe obstructive physiology on PFTs (FEV1/FVC <0.70 and FEV1 < 50% normal), if done.

     21. Subjects who have an active infection requiring systemic antibiotics or an elevated white blood count (above the local laboratory reference ranges).

     22. Have a history of active drug addiction, active alcohol abuse, or psychiatric hospital admission for psychosis within the prior 2 years.

     23. Are currently participating in a clinical study or investigation. 24. Subject otherwise not appropriate for study as determined by the investigator and subjects who are unwilling to comply with the study protocol, or subjects with a history of non-compliance. The reasons must be documented.

     25. Subjects contraindicated for trans-septal puncture, TEE or ICE.

   Intra Procedural Exclusion Criteria:

   (Intra Procedural Exclusion Criteria will be determined immediately after intracardiac echocardiography or transesophageal echocardiography determination of left atrial anatomy and just before transseptal puncture) 26. Anatomical anomaly on TEE or ICE that precludes implantation of the V-LAPIM across the interatrial septum (Fossa Ovalis) including: Septal thickness at fossa > 5 mm, FO Dimension <16mm, ASD or PFO with more than a trace amount of shunting, intra-cardiac thrombus felt to be acute and not present on prior exams and abnormal septum, e.g., a hypermobile septum or a septal aneurysm.

   27. Inadequate vascular access for implantation of V-LAPIM or are unable to tolerate a right heart catheterization (RHC).

   28. Severe pulmonary hypertension at index procedure above 70 mmHg or PVR at index procedure above 4.0 Woods Units (mmHg L-1 min-1), while these cannot be lowered with vasodilators.

   29. Resting systolic Blood Pressure <90 or >180 mmHg, not corrected with IV fluid administration or vasodilators.

Ages: 22 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
LAP measurement | Up to 12 months post-procedure
  Freedom from failure of the V-LAP system to obtain LAP measurement from the sensor implant and transmit the LAP data to the V-LAPDD Data Display and the V-LAPPSM Patient Guidance Application.
Safety Endpoint - Major Adverse Cardiac and Neurological Events (MACNE) | Up to three months post-procedure
  Number of participants with study (Device and/ or system) related to Major Adverse Cardiac and Neurological Events (MACNE) - as defined in the protocol, as by the independent Clinical Events Committee
Performance accuracy | At index (Implantation visit)
  LAP accuracy validation, concordance of the V-LAP implant measurement with pulmonary capillary wedge pressure (PCWP) measurement

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Bayés-Genís, MD PhD, Principal Investigator — Universitari Germans Trias i Pujol in Badalona; David Meerkin, MD, Principal Investigator — Shaare Zedek Medical Center Jerusalem, Israel; Ran Kornowski, MD PhD, Principal Investigator — Rabin Belinson, Medical Center - Israel; Filippo Crea, MD PhD, Principal Investigator — Universitario Agostino Gemelli
Locations (1):
- Rabin Belinson, Medical Center - Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No